CLINICAL TRIAL: NCT05915819
Title: Comparative Effects of Plyometric Training and Eccentric Muscle Training on Functional Performance in Weightlifters
Brief Title: Effects of Plyometric Training and Eccentric Muscle Training on Functional Performance in Weightlifters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/RCR&AHS/23/0419
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Functional Performance
Keywords: adult; connective Tissue; lifting; plyometric exercises; signal transduction
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Experimental): This group will trained with Plyometric training This training of this group will be Plyometric in which many exercises of both region upper extremity and lower extremity guided to weightlifter for assessment of functional performance. Before starting the plyometric training the trainer will perform a traditional exercise like push-ups or cycling for warmup, 5-10minutes. In plyometric training the exercise we will focus all over the body fitness, The exercise prescription according to weeks, sets and repetition.
  sessions will be 6 days a week 6 weeks training sessions
  Interventions: Other: Plyometric Training
- Eccentric Training (Experimental): This group will Trained with Eccentric muscle training Before starting the eccentric heavy load exercise trainers will perform warm up exercise then we will continue training.
  Sessions will be 6 days a week 6 weeks training sessions
  Interventions: Other: Eccentric Training

INTERVENTIONS:
Other: Plyometric Training — Exercise prescription according to weeks, sets and repetition. Weeks 1 and 2 1-2 sets / 10 repetitions Double leg jump Medicine ball(MB) stuffer flutter MB overhead throw MB single leg dip, Arrow cone drill Figure 8 drill Weeks 3 and 4 1-2 sets / 8 repetitions Ankle jumps Lateral cone hops Zigzag jump drill MB chest pass Jump & turn 90° High-5 drill MB split squat Power skipping Clock drill T-drill Weeks 5 and 6 1-2 sets / 6 repetitions Dot drill Single leg cone hops Long jump and sprint Single leg zigzag drill MB lunge chest pass Jump and turn 180° Split squat jump Alternate bounding X-drill Shuttle drill
  Arms: Plyometric Training
Other: Eccentric Training — The eccentric training will be Pull-ups 3-5 sets X 6-8 reps Glute-ham raise 3-5 sets x 10rep Manual glute-ham raise 3-5 sets x 10rep single-leg Romanian dead lift or good morning(barbell or dumbbell) 3-5 sets x 10rep Glute-bridge and hip thrust (can also perform single leg movement) 3-5 sets x 10rep Half-kneel-bottom-up press-eccentric only. 3-5 sets x 8rep The eccentric exercise technique will be 2/1 technique, Two-movement technique, Slow/super slow, Negative (supramax)
  Arms: Eccentric Training

SUMMARY:
Stretching, pressing, and lifting large weights with speed and balance all require strong muscles. In plyometric exercise, the same muscle must be stretched and rapidly contracted in order to make quick, strong motions. Plyometric exercises include explosive jumps, hops, bounds, and skips. A major component in becoming a better weight lifter is plyometric training that focuses on the lower limb. Additionally, as the muscle produces and stores kinetic energy, it is crucial to increase muscle power, strength, and endurance. Eccentric muscular activity relate to the dynamic extension of muscle tissue in resistance to an external force or load. Eccentric muscular activities have been demonstrated to induce a higher elevation of molecular signalling pathways connected to muscle and connective tissue anabolism and increased activation of satellite cells.

This study will be a Randomized control trial and occur on improving functional performance in weightlifters. The inclusion criteria are, training will perform only elite weightlifters, aged between 20-30 years, and have 4-5 years of weightlifting experience. In this study we will compare two groups including 20 participants, 10 participants will be trained in plyometric exercises and 10 participants will be on eccentric muscle training and we will analyze which group will enhance functional performance. We will use an Assessment scale to assess the upper and lower extremity dysfunction through the Upper extremity assessment scale and Lower extremity assessment scale.

DETAILED DESCRIPTION:
To compare the effect of plyometrics training and eccentric muscle training to improve functional performance in weightlifters.

The study will be Randomized control trial. Non-Probablity propulsive techninque DATA COLLECTION TOOLS Lower Extremity Functional Scale Upper extremity Functional scale Vertical jump & long jump Seated medicine Ball toss V-sit and reach test The Data will be analyzed using SPSS for windows software version 25. Statistical significance P=0.05. After assessing the normality of current data by shapiro wilk test. it will be decided whether parametric or non parametric test will be used within the groups or between 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Elite competitive weightlifters
* Age 20-30 year
* Weightlifting experience 4-5 years
* The weightlifter can perform all functional activities

Exclusion Criteria:

* female
* Low BMI
* History of injury,
* History of surgery and pain

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
Lower extremity functional scale | 6 weeks
  A reliable patient-rated outcome measure (PROM) for assessing lower extremity function is the lower extremity functional scale (LEFS). For a variety of lower-extremity diseases, the Lower Extremity Functional Scale (LEFS) is used to assess "patients' initial function, ongoing improvement, and outcome
Upper extremity Functional scale | 6 weeks
  A patient-reported outcome measure called the upper Extremity Functional scale is used to evaluate functional impairment in people with musculoskeletal upper limb dysfunction.
Vertical jump & long jump | 6 weeks
  Subjects were instructed to jump as high as possible and touch the highest point. The vertical jump was calculated by subtracting a subject's standing reach height from his maximal jump height.
  The standing long jump is measure on a mat which was fixed to the floor. Subjects were permitted to perform a countermovement prior to jumping vertically or horizontally Subjects were instructed to jump as high as possible and touch the highest point. The vertical jump was calculated by subtracting a subject's standing reach height from his maximal jump height.
  The standing long jump is measure on a mat which was fixed to the floor. Subjects were permitted to perform a countermovement prior to jumping vertically or horizontally
Seated medicine Ball toss | 6 weeks
  The seated medicine ball toss is to perform with a 3.6 kg medicine ball. The participants sat on the floor with their back against a wall and were instructed to toss the ball as far as they could with both hands at an approximate angle of 45° (similar to a chest pass). Prior to each toss the ball with weightlifting chalk so that when the ball landed on the floor it left a distinctive mark that allowed for a precise measurement. The distance from the wall to the near edge of the mark on the floor made by the ball was measured
V-sit and reach test | 6 weeks
  V-sit and reach test is use to measure flexibility of back muscles or hamstring muscles in a temperature control environment.1) Mark a baseline on the floor. 2) A ruler is placed perpendicularly to the baseline which cross the baseline at 15inches. 3) Sit with the heels on the baseline with feet 12inches apart. 4) With the legs straight, slowly bends forward to reach the furthest point of the ruler. 5) Hold for 2 seconds and record the distance. 6) Perform three trials with the best score recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nosheen Manzoor, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Hajvery sports complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serrano BA. Rotator Cuff Pathology in Olympic Weightlifting: A Comprehensive Review of Incidence, Diagnosis, Management, and Rehabilitation. 2020.
- [Background] Riemann BL, Mercado M, Erickson K, Grosicki GJ. Comparison of balance performance between masters Olympic weightlifters and runners. Scand J Med Sci Sports. 2020 Sep;30(9):1586-1593. doi: 10.1111/sms.13729. Epub 2020 Jun 22. PMID 32474974
- [Background] Gharib S. Effect of functional strength training on snatch performance for weightlifters. Turkish Journal of Kinesiology. 2018;4(2):47-52
- [Background] Berton R, Lixandrao ME, Pinto E Silva CM, Tricoli V. Effects of weightlifting exercise, traditional resistance and plyometric training on countermovement jump performance: a meta-analysis. J Sports Sci. 2018 Sep;36(18):2038-2044. doi: 10.1080/02640414.2018.1434746. Epub 2018 Feb 1. PMID 29385904
- [Background] Fischetti F, Vilardi A, Cataldi S, Greco G. Effects of plyometric training program on speed and explosive strength of lower limbs in young athletes. Journal of Physical Education & Sport. 2018;18(4)
- [Background] Hu J, Zulkapri IB. Analysis of Physical Fitness Evaluation System for Weightlifters Based on Analytic Hierarchy Process. Mobile Information Systems. 2022;2022
- [Background] Kipp K. IDENTIFYING JOINT-SPECIFIC LIMITATIONS AND TARGETS FOR IMPROVING WEIGHTLIFTING PERFORMANCE. ISBS Proceedings Archive. 2021;39(1):200.
- [Background] Suchomel TJ, Wagle JP, Douglas J, Taber CB, Harden M, Haff GG, Stone MH. Implementing Eccentric Resistance Training-Part 1: A Brief Review of Existing Methods. J Funct Morphol Kinesiol. 2019 Jun 24;4(2):38. doi: 10.3390/jfmk4020038. PMID 33467353
- [Background] Morris SJ, Oliver JL, Pedley JS, Haff GG, Lloyd RS. Comparison of Weightlifting, Traditional Resistance Training and Plyometrics on Strength, Power and Speed: A Systematic Review with Meta-Analysis. Sports Med. 2022 Jul;52(7):1533-1554. doi: 10.1007/s40279-021-01627-2. Epub 2022 Jan 13. PMID 35025093
- [Background] Hawkins SB, Doyle TL, McGuigan MR. The effect of different training programs on eccentric energy utilization in college-aged males. J Strength Cond Res. 2009 Oct;23(7):1996-2002. doi: 10.1519/JSC.0b013e3181b3dd57. PMID 19855323
- [Background] Hammami R, Duncan MJ, Nebigh A, Werfelli H, Rebai H. The Effects of 6 Weeks Eccentric Training on Speed, Dynamic Balance, Muscle Strength, Power, and Lower Limb Asymmetry in Prepubescent Weightlifters. J Strength Cond Res. 2022 Apr 1;36(4):955-962. doi: 10.1519/JSC.0000000000003598. PMID 32483061
- [Background] di Cagno A, Iuliano E, Buonsenso A, Giombini A, Di Martino G, Parisi A, Calcagno G, Fiorilli G. Effects of Accentuated Eccentric Training vs Plyometric Training on Performance of Young Elite Fencers. J Sports Sci Med. 2020 Nov 19;19(4):703-713. eCollection 2020 Dec. PMID 33239944
- [Background] Grgic J, Schoenfeld BJ, Mikulic P. Effects of plyometric vs. resistance training on skeletal muscle hypertrophy: A review. J Sport Health Sci. 2021 Sep;10(5):530-536. doi: 10.1016/j.jshs.2020.06.010. Epub 2020 Jun 21. PMID 32579911
- [Background] Kipp K, Harris C, Sabick MB. Lower extremity biomechanics during weightlifting exercise vary across joint and load. J Strength Cond Res. 2011 May;25(5):1229-34. doi: 10.1519/JSC.0b013e3181da780b. PMID 21240030
- [Background] Alawna M, Mohamed AA. Short-term and long-term effects of ankle joint taping and bandaging on balance, proprioception and vertical jump among volleyball players with chronic ankle instability. Phys Ther Sport. 2020 Nov;46:145-154. doi: 10.1016/j.ptsp.2020.08.015. Epub 2020 Aug 29. PMID 32937273
- [Background] Cacchio A, De Blasis E, Necozione S, Rosa F, Riddle DL, di Orio F, De Blasis D, Santilli V. The Italian version of the lower extremity functional scale was reliable, valid, and responsive. J Clin Epidemiol. 2010 May;63(5):550-7. doi: 10.1016/j.jclinepi.2009.08.001. Epub 2009 Nov 12. PMID 19913388
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Chesworth BM, Hamilton CB, Walton DM, Benoit M, Blake TA, Bredy H, Burns C, Chan L, Frey E, Gillies G, Gravelle T, Ho R, Holmes R, Lavallee RL, MacKinnon M, Merchant AJ, Sherman T, Spears K, Yardley D. Reliability and validity of two versions of the upper extremity functional index. Physiother Can. 2014 Summer;66(3):243-53. doi: 10.3138/ptc.2013-45. PMID 25125777
- [Background] Faigenbaum AD, McFarland JE, Keiper FB, Tevlin W, Ratamess NA, Kang J, Hoffman JR. Effects of a short-term plyometric and resistance training program on fitness performance in boys age 12 to 15 years. J Sports Sci Med. 2007 Dec 1;6(4):519-25. eCollection 2007. PMID 24149486
- [Background] Amiri-Khorasani M, Kellis E. Acute Effects of Different Agonist and Antagonist Stretching Arrangements on Static and Dynamic Range of Motion. Asian J Sports Med. 2015 Dec;6(4):e26844. doi: 10.5812/asjsm.26844. Epub 2015 Dec 1. PMID 26715975
- [Background] Attrey P, Yadav M, Singh S, IP, R TD, Yamunanagar H. RELATIONSHIP BETWEEN PASSIVE STRAIGHT LEG RAISING TEST AND V-SIT AND REACH TEST IN MEASURING THE HAMSTRING FLEXIBILITY. Journal DOI. 2016:44975451
- [Background] Mike J, Kerksick CM, Kravitz L. How to incorporate eccentric training into a resistance training program. Strength & Conditioning Journal. 2015;37(1):5-17.